CLINICAL TRIAL: NCT00655538
Title: A Randomized, Placebo-controlled Study of the Safety, Tolerability and Effect on Endothelial Function, as Measured by Flow Mediated Dilatation, of RO4607381 in Patients With Coronary Heart Disease (CHD) or CHD Risk Equivalents.
Brief Title: A Study Assessing the Effect of RO4607381 on Vascular Function in Patients With Coronary Heart Disease (CHD) or CHD-Risk Equivalent Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC21144; 2007-003406-10
Record Dates: First submitted 2008-03-28; First posted 2008-04-10 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dalcetrapib (Experimental)
  Interventions: Drug: dalcetrapib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — po daily for 36 weeks
  Arms: Placebo
Drug: dalcetrapib — 600mg po daily for 36 weeks
  Arms: Dalcetrapib

SUMMARY:
This study will assess the safety, tolerability and efficacy of RO4607381 in patients with coronary heart disease (CHD) or CHD risk equivalents. Patients will be randomized to receive either RO4607381 600mg po daily or placebo po daily. Endothelial function will be measured by flow mediated dilatation and blood pressure monitoring will be assessed. The anticipated time on study treatment is up to 12 months, and the target sample size is up to 500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* CHD or CHD risk equivalent;
* appropriately treated for accepted LDL-C level.

Exclusion Criteria:

* treatment with drugs raising HDL-C (eg niacin, fibrates);
* uncontrolled hypertension;
* recent (within 3 months) clinically significant coronary events, transient ischemic attacks or cerebrovascular accident;
* severe anemia;
* poorly controlled diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- Feldkirch, Austria
- Paris, France
- Germany (5):
  - Bonn
  - Dortmund
  - Frankfurt
  - Mainz
  - Wuppertal
- Pisa, Tuscany, Italy
- Netherlands (12):
  - Amsterdam
  - Breda
  - Eindhoven
  - Goes
  - Groningen
  - Hoorn
  - Leiderdorp
  - Nijmegen
  - Rotterdam
  - Utrecht
  - Velp
  - Zoetermeer
- Switzerland (2):
  - Lugano
  - Zurich
- Cardiff, United Kingdom

REFERENCES:
- [Derived] Luscher TF, Taddei S, Kaski JC, Jukema JW, Kallend D, Munzel T, Kastelein JJ, Deanfield JE; dal-VESSEL Investigators. Vascular effects and safety of dalcetrapib in patients with or at risk of coronary heart disease: the dal-VESSEL randomized clinical trial. Eur Heart J. 2012 Apr;33(7):857-65. doi: 10.1093/eurheartj/ehs019. Epub 2012 Feb 16. PMID 22345126
- [Derived] Kastelein JJ, Duivenvoorden R, Deanfield J, de Groot E, Jukema JW, Kaski JC, Munzel T, Taddei S, Lehnert V, Burgess T, Kallend D, Luscher TF. Rationale and design of dal-VESSEL: a study to assess the safety and efficacy of dalcetrapib on endothelial function using brachial artery flow-mediated vasodilatation. Curr Med Res Opin. 2011 Jan;27(1):141-50. doi: 10.1185/03007995.2010.536207. Epub 2010 Dec 6. PMID 21128879

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalcetrapib | Placebo
Started | 238 | 238
Completed | 214 | 211
Not Completed | 24 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalcetrapib | Placebo | Total
Number analyzed (Participants) | 232 | 234 | 466
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (7.05) | 61.9 (7.92) | 62.1 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 211 | 422
  Male | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in % Flow Mediated Dilatation (FMD)
Time Frame: Baseline and 12 weeks
Population: 10 subjects dropped before week 12
Measure: Least Squares Mean (Standard Error); unit: %FMD
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 232 | 234
%FMD | 0.09 (0.13) | 0.32 (0.13)

2. Primary Outcome: Change From Baseline in Mean BP, Measured by BP Monitoring
Time Frame: Baseline and 4 weeks
Population: not all participants were tested
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 235 | 237
mmHg | 0.91 (0.57) | 0.31 (0.57)

3. Secondary Outcome: Change From Baseline in % FMD
Time Frame: baseline and 36 weeks
Population: not all participants were tested
Measure: Least Squares Mean (Standard Deviation); unit: %FMD
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 232 | 234
%FMD | 10.50 (6.27) | 20.13 (5.95)

4. Secondary Outcome: Percent Change in HDL-C, LDL-C, Total Cholesterol, Triglycerides, ApoA1, ApoB
Time Frame: Baseline to 36 weeks
Population: not all participants were tested
Measure: Least Squares Mean (Standard Error); unit: Percent change in mg/dL
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 207 | 211
Percent change in mg/dL
  HDL-C | 30.70 (1.45) | -0.14 (1.42)
  LDL-C | 4.43 (2.22) | 8.72 (2.18)
  Total Cholesterol | 8.66 (1.20) | 5.90 (1.18)
  Triglycerides | -2.58 (2.66) | 11.62 (2.61)
  ApoA1 | 12.84 (0.97) | 2.61 (0.96)
  ApoB | -2.70 (1.23) | 1.98 (1.21)

5. Secondary Outcome: CETP Activity
Time Frame: Up to 36 weeks
Population: not all participants were tested
Measure: Least Squares Mean (Standard Error); unit: Percent change pMOL/uL/hr
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 207 | 210
Percent change pMOL/uL/hr | -48.66 (2.12) | 7.37 (2.09)

6. Secondary Outcome: Percent Change From Baseline of sP-Selectin, sE-Selectin, Soluble Intracellular Adhesion Molecule, Soluble Vascular Cell Molecule, Lipoprotein-associated phospholipaseA2s, Matrix Metalloproteinase-3, Matrix metalloproteinase9
Time Frame: Baseline and 36 weeks
Population: not all participants were tested
Measure: Mean (Standard Error); unit: Percent change in ng/mL
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 207 | 211
Percent change in ng/mL
  sP-Selectin | -1.83 (1.58) | 0.24 (1.54)
  sE-Selectin | 6.01 (1.95) | 6.08 (1.90)
  Soluble intracellular adhesion molecule | 1.05 (0.95) | 2.01 (0.94)
  Soluble vascular cell molecule | 3.60 (0.79) | 1.86 (0.78)
  Lipoprotein-associated phospholipaseA2s | 23.24 (3.34) | 5.80 (3.29)
  Matrix metalloproteinase-3 | 3.46 (2.12) | 3.44 (2.07)
  Matrix metalloproteinase9 | 28.12 (10.97) | 20.36 (10.75)

7. Secondary Outcome: Change From Baseline in Mean BP, Measured by BP Monitoring
Time Frame: Up to 36 weeks
Population: not all participants were tested
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 235 | 237
mmHg | 1.93 (0.60) | 1.17 (0.59)

8. Secondary Outcome: Percent Change CETP Mass
Time Frame: baseline to 36 weeks
Population: not all participants were tested
Measure: Least Squares Mean (Standard Error); unit: Percent change in ug/mL
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 207 | 211
Percent change in ug/mL | 94.19 (2.70) | 5.17 (2.65)

ADVERSE EVENTS:
Arm/Group | Dalcetrapib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/236 | 1/236
Serious Adverse Events (participants affected / at risk) | 12/236 | 14/236
Other Adverse Events (participants affected / at risk) | 92/236 | 112/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalcetrapib (N=236) | Placebo (N=236)
Angina Pectoris (Cardiac disorders) | 1 | 2
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial Fibrilation (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Appendicitis Perforated (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0
Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Migrane (Nervous system disorders) | 0 | 1
Transient Ischemic Attack (Nervous system disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Purexia (General disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urethral Stenosis (Renal and urinary disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Gastric Disorder (Gastrointestinal disorders) | 1 | 0
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dalcetrapib (N=236) | Placebo (N=236)
Nasopharyngitis (Infections and infestations) | 38 | 42
Influenza (Infections and infestations) | 9 | 15
Diarrhea (Gastrointestinal disorders) | 27 | 26
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 16
Headache (Nervous system disorders) | 10 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No